CLINICAL TRIAL: NCT01520961
Title: Approach Your Neck Fracture
Brief Title: Functional Recovery After Partial Hip Arthroplasty: Anterior or Posterolateral Approach?
Acronym: AYNF
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician Responsible of Clinical Research, Hospital Ambroise Paré Paris
Other Study IDs: APR122011
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Hip Arthroplasty; Femoral Neck Fractures
Keywords: Partial Hip Arthroplasty
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hueter Anterior Approach
- posterolateral approach

SUMMARY:
Hueter anterior approach as described by Siguier allows an anatomical approach without muscle or tendon sections. It minimizes the rate of dislocation after primary total hip arthroplasty (1.5%, Sariali)and seems to allow quicker rehabilitation.

The investigators hypothesis was Hueter anterior approach allows quicker functional recovery after partial hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Femoral Neck Fracture
* Partial Hip Arthroplasty

Exclusion Criteria:

* Total Hip Arthroplasty
* Osteosynthesis
* Pathologic fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Partial Hip Arthroplasty for Femoral Neck Fracture
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Measurement of mobility | Timed Get Up and Go Test at six weeks
  Efficacity issue

SECONDARY OUTCOMES:
Measurement of mobility | Using 2 cruches or walker at 6 weeks after surgery
Dislocation rate | At 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ambroise Paré Hospital. Orthopaedic surgery department, Boulogne-Billancourt, Île-de-France Region, France